CLINICAL TRIAL: NCT00003329
Title: ECOG Laboratory Study: Mapping Interactive Cancer Susceptibility Loci
Brief Title: Identification of Genes Associated With Cancer in Patients and Siblings Who Have Cancer
Status: Completed | Type: Observational
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000066283; U10CA021115 (NIH); ECOG-1Y97
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer; Colorectal Cancer; Lung Cancer; Prostate Cancer
Keywords: stage I colon cancer; stage II colon cancer; stage III colon cancer; stage IV colon cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage III non-small cell lung cancer; limited stage small cell lung cancer; extensive stage small cell lung cancer; stage I prostate cancer; stage II prostate cancer; stage III prostate cancer; stage IV prostate cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Lung Neoplasms; Prostatic Neoplasms; Colonic Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Chromosome Mapping

INTERVENTIONS:
Genetic: gene mapping

SUMMARY:
RATIONALE: Identification of genes that may be associated with developing certain types of cancer may someday provide important information about a person's risk of getting cancer.

PURPOSE: This clinical trial is studying to see if certain genes may be associated with cancer in patients with cancer of the breast, prostate, lung, or colon and siblings of these patients.

DETAILED DESCRIPTION:
OBJECTIVES:

* Gather allele-sharing statistics at approximately 100 candidate loci throughout the human genome most likely to influence genetic risk of cancer.
* Use these allele-sharing statistics to test the interaction of each locus individually with cancer-associated, rare alleles of HRAS1.
* Generalize this approach for one of four cancers (breast, colon, lung, or prostate), using allele-sharing statistics to test the interaction of each locus with every other locus.
* Replicate positive results in a distinct set of sibling pairs with cancer.
* Examine, when loci contributing to risk are detected, the influence of this genetic background on clinical outcomes, such as survival.

OUTLINE: Each patient-sibling pair completes a family history questionnaire about the incidence of cancer in the family. Blood samples are obtained from both the patient and the sibling (and both living parents, if available).

The blood samples are genotyped using approximately 300 micro-satellite markers flanking 100 candidate genes previously implicated in genetic risk for cancer. Certain loci are a priority due to their association with HRAS1: BRCA1 and all known mismatch repair loci; other repair genes, such as ATM; the Bloom's syndrome locus; and the XRCC group. Other genes are also mapped.

Patients do not receive the results of the genetic testing and the results do not influence the type and duration of treatment.

Patients only are followed annually.

PROJECTED ACCRUAL: This study will accrue 1,000 patient-sibling pairs for breast cancer. After 18 months, another 1,000 patient-sibling pairs will be accrued for breast cancer. Therefore, up to 2,000 patient-sibling pairs will be accrued over 5 years. (Feasibility of accruing pairs for lung, colon, and prostate cancer is being assessed.)

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed colon, lung, prostate, or invasive breast cancer

  * No ductal or lobular carcinoma in situ of the breast only
* Patient and natural full sibling must have (or have had) cancer of the same type
* Participants in E-3Y92 not eligible
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* Not specified

Menopausal status:

* Not specified

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Ages: 0 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 1998-04-07 (Actual); Primary Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (32):
- United States (32):
  - Lucy Curci Cancer Center at Eisenhower Memorial Hospital and Medical Center, Rancho Mirage, California
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Eugene M. and Christine E. Lynn Cancer Institute at Boca Raton Community Hospital, Boca Raton, Florida
  - Lakeland Regional Cancer Center at Lakeland Regional Medical Center, Lakeland, Florida
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago Westside Hospital, Chicago, Illinois
  - Evanston Northwestern Healthcare - Evanston Hospital, Evanston, Illinois
  - Hematology Oncology Associates - Skokie, Skokie, Illinois
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - Finger Lakes Hematology and Oncology, Clifton Springs, New York
  - Our Lady of Mercy Medical Center Comprehensive Cancer Center, The Bronx, New York
  - Joan Karnell Cancer Center at Pennsylvania Hospital, Philadelphia, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - Jennersville Regional Hospital, West Grove, Pennsylvania
  - Fox Valley Hematology and Oncology - East Grant Street, Appleton, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - All Saints Cancer Center at Wheaton Franciscan Healthcare, Racine, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin

REFERENCES:
- [Result] Larson GP, Ding Y, Cheng LS, Lundberg C, Gagalang V, Rivas G, Geller L, Weitzel J, MacDonald D, Archambeau J, Slater J, Neuberg D, Daly MB, Angel I, Benson AB 3rd, Smith K, Kirkwood JM, O'Dwyer PJ, Raskay B, Sutphen R, Drew R, Stewart JA, Werndli J, Johnson D, Ruckdeschel JC, Elston RC, Krontiris TG. Genetic linkage of prostate cancer risk to the chromosome 3 region bearing FHIT. Cancer Res. 2005 Feb 1;65(3):805-14. PMID 15705877
- [Result] Krontiris TG, Larson M, Weitzel JN, et al.: Mapping interactive cancer susceptibility loci: Eastern Cooperative Oncology Group. [Abstract] Proceedings of the American Society of Clinical Oncology 17: A2147, 560a, 1998.